CLINICAL TRIAL: NCT07108790
Title: Comparative Study Between Bovine Bone With or Without Concentrated Growth Factor in the Treatment of Chronic Periodontitis
Brief Title: Bovine Bone With or Without Concentrated Growth Factor in the Treatment of Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nouran Elsayed Elbadawy, B.D.S of Oral Medicine, Periodontology, Oral Diagnosis & Oral Radiology, Faculty of Dentistry, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-OMPDR-3-22-11
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Bovine Bone; Concentrated Growth Factor; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ι (Experimental): Ten sites were treated by concentrated growth factors (CGF), collagen membrane, and xenograft bone graft.
  Interventions: Other: Concentrated growth factors, collagen membrane and xenograft bone graft
- Group ΙΙ (Active Comparator): Ten sites were treated with a collagen membrane and a xenograft bone graft.
  Interventions: Other: Collagen membrane and xenograft bone graft

INTERVENTIONS:
Other: Concentrated growth factors, collagen membrane and xenograft bone graft — Ten sites were treated by concentrated growth factors (CGF), collagen membrane, and xenograft bone graft.
  Arms: Group Ι
Other: Collagen membrane and xenograft bone graft — Ten sites were treated with a collagen membrane and a xenograft bone graft.
  Arms: Group ΙΙ

SUMMARY:
The aim of this study is to compare bovine bone with or without concentrated growth factor in the treatment of chronic periodontitis.

DETAILED DESCRIPTION:
Periodontitis is an infection-driven inflammatory disease resulting from dental plaque accumulation at the gingival margin, triggering an inflammatory response that leads to microbial alterations and may have severe consequences for the periodontium of susceptible individuals.

The xenograft most commonly used in periodontal regeneration procedures is the deproteinized bovine or equine bone mineral.

Platelets are known to play a significant role in guided tissue regeneration (GTR) by releasing several growth factors, such as platelet-derived growth factor (PDGF), and plasma rich in growth factors (PRGF), which are present in platelet-rich plasma (PRP), a first-generation platelet concentrate. Platelet-rich fibrin (PRF) and concentrated growth factors (CGF) are considered the second generation of platelet concentrate.

ELIGIBILITY:
Inclusion Criteria:

* Presence of angular periodontal intra-bony defects with a pocket depth (PD) ≥ 5mm.
* Optimal compliance as evidenced by no missed treatment appointments and a positive attitude towards oral hygiene.
* Full-mouth bleeding score ≤ 25%.

Exclusion Criteria:

* Patients with relevant medical conditions that may affect periodontal regeneration and periodontal surgery.
* Patients who have any disease or take any medication that affects the normal number or function of platelets.
* Smokers.
* Pregnant or lactating women.
* Patients in whom periodontal surgery had previously been carried out on the selected site.
* Patients with aggressive periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Probing Pocket depth | 6 months post-procedure
  Probing Pocket depth (PPD) was measured.

SECONDARY OUTCOMES:
Clinical attachment level | 6 months post-procedure
  Clinical attachment level (CAL) was measured.
Bleeding on probing | 6 months post-procedure
  Bleeding on probing (BOP) was measured.
Plaque index | 6 months post-procedure
  Plaque index (PI) was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.